CLINICAL TRIAL: NCT07093697
Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW5121 Compared to DW51211 and DW51212
Brief Title: A Study to Evaluate the Efficacy and Safety of DW5121 Compared to DW51211 and DW51212
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW5121-302
Record Dates: First submitted 2025-06-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Acute Bronchitis
Keywords: Acute bronchitis; Bronchitis Severity Score; respiratory infection; Phase 3 clinical trial
MeSH Terms: conditions — Bronchitis; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DW5121 Group (Experimental): Participants receive DW5121, 2 tablets orally, DW51211 Placebo, 2 tablets orally, DW51212 Placebo, 1 tablets orally, 3 times a day after meals for 7 days
  Interventions: Drug: DW5121
- DW51211 Control Group (Active Comparator): Participants receive DW5121 placebo, 2 tablets orally, DW51211, 2 tablets orally, DW51212 Placebo, 1 tablets orally, 3 times a day after meals for 7 days
  Interventions: Drug: DW51211
- DW51212 Control Group (Active Comparator): Participants receive DW5121 placebo, 2 tablets orally, DW51211 placebo, 2 tablets orally, DW51212 , 1 tablets orally, 3 times a day after meals for 7 days
  Interventions: Drug: DW51212

INTERVENTIONS:
Drug: DW5121 — Participants receive DW5121, 2 tablets orally, DW51211 Placebo, 2 tablets orally, DW51212 Placebo, 1 tablets orally, 3 times a day after meals for 7 days
  Arms: DW5121 Group
Drug: DW51211 — Participants receive DW5121 placebo, 2 tablets orally, DW51211, 2 tablets orally, DW51212 Placebo, 1 tablets orally, 3 times a day after meals for 7 days
  Arms: DW51211 Control Group
Drug: DW51212 — Participants receive DW5121 placebo, 2 tablets orally, DW51211 placebo, 2 tablets orally, DW51212 , 1 tablets orally, 3 times a day after meals for 7 days
  Arms: DW51212 Control Group

SUMMARY:
This is a Phase 3, randomized, double-blind, active-controlled, parallel-group, multi-center clinical trial to evaluate the efficacy and safety of DW5121 compared to DW51211 and DW51212 in patients with acute bronchitis. The primary objective is to demonstrate the superiority of DW5121 over DW51211 and DW51212 by comparing the change in total Bronchitis Severity Score (BSS) at Day 4 after administration. Approximately equal numbers of patients were randomized in a 1:1:1 ratio to receive DW5121, DW51211, or DW51212 for 7 days. Efficacy and safety assessments were conducted at Day 4 and Day 7, with a follow-up contact approximately 5 days after the end of treatment to monitor adverse events.

DETAILED DESCRIPTION:
Acute bronchitis is a common respiratory condition characterized by inflammation of the bronchial tubes, leading to symptoms such as coughing, sputum production, and discomfort. Effective treatment options with improved symptom control and safety profiles are needed.

This Phase 3, randomized, double-blind, parallel-group, multi-center, active-controlled, superiority trial aims to evaluate the efficacy and safety of DW5121 compared to DW51211 and DW51212 in patients with acute bronchitis. Eligible participants were randomized in a 1:1:1 ratio to receive either DW5121, DW51211, or DW51212 for 7 days.

The primary objective is to assess the change in total Bronchitis Severity Score (BSS) at Day 4 (±1 day) after drug administration, and to demonstrate the superiority of DW5121 compared to both comparators.

The secondary objectives include:

1. Comparison of BSS score changes at Day 4 between DW5121 and each comparator, including statistical significance.
2. Evaluation of overall efficacy and safety of DW5121 relative to DW51211 and DW51212.

Participants visited the study site at baseline, Day 4 (Visit 3), and Day 7 (Visit 4). A follow-up safety check (Visit 5) was conducted approximately 5 days after the last visit. Additional site visits or assessments were performed as necessary based on investigator's discretion to monitor adverse events.

This study provides important data on the potential benefits of DW5121 in managing symptoms of acute bronchitis, with an emphasis on both clinical efficacy and patient safety.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Male or female aged ≥19 years and <80 years at the time of informed consent.
2. Patients diagnosed with acute bronchitis with productive cough symptoms within 48 hours prior to randomization (diagnosis based on clinical symptoms and chest X-ray; additional bacterial or viral testing may be performed if necessary).
3. Subjects with a total Bronchitis Severity Score (BSS) of ≥5 and a sputum score of at least 1 at the randomization visit.
4. Subjects who voluntarily provided written informed consent to participate in this clinical trial.

Exclusion Criteria:

Subjects who meet any of the following conditions will not be eligible to participate in this clinical trial:

1. History of hypersensitivity to any component of the investigational product or to drugs of a similar class.

2. Presence of any of the following medical histories or past surgical/interventional histories:

1. Active infections requiring systemic antibiotic therapy
2. Severe pulmonary diseases as determined by the investigator (e.g., bronchiectasis, bronchogenic carcinoma, interstitial lung disease, pneumonia, active tuberculosis, cystic fibrosis, chronic obstructive pulmonary disease, asthma, chronic bronchitis, emphysema, etc.) or clinically significant abnormal findings on chest X-ray
3. Obstructive sleep apnea syndrome
4. Glaucoma or elevated intraocular pressure
5. Lower urinary tract obstruction (e.g., benign prostatic hyperplasia) or voiding dysfunction
6. Hemorrhagic diathesis or bleeding tendency
7. Hepatic dysfunction (ALT or AST > 3 × upper limit of normal)
8. Renal impairment (glomerular filtration rate < 30 mL/min)

   *eGFR (mL/min/1.73m²) = 175 × (serum creatinine)^(-1.154) × (age)^(-0.203) × 0.742 (if female)
9. Uncontrolled thyroid dysfunction (TSH ≥ 1.5 × ULN)
10. Uncontrolled diabetes mellitus (HbA1c > 9.0%)
11. Uncontrolled hypertension (systolic or diastolic blood pressure ≥ 160/100 mmHg)
12. Significant cardiovascular diseases as determined by the investigator (e.g., heart failure of NYHA class III/IV, atherosclerosis, pulmonary hypertension, peripheral artery disease) or QTc interval > 450 msec or other clinically significant ECG abnormalities
13. Active peptic ulcer, gastrointestinal bleeding, or pyloroduodenal obstruction
14. Central nervous system diseases such as epilepsy
15. Subjects with rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
16. History of malignancy except in the following cases:

(1) Disease-free for at least 5 years following completion of cancer treatment

(2) Subjects who have completed curative resection of basal cell carcinoma or squamous cell carcinoma of the skin, curative surgery for papillary thyroid carcinoma, or successful treatment of cervical carcinoma in situ at least 3 years prior to screening

3. Subjects expected to require any of the following medications during the clinical trial:

1. Antibiotics, antivirals, systemic/inhaled glucocorticosteroids
2. ACE inhibitors or ARBs (Note: Subjects on long-term stable doses of ACEIs or ARBs may be included)
3. Mucolytics, expectorants, antitussives, herbal medicines with antitussive/expectorant effects
4. Leukotriene receptor antagonists, antihistamines, β2 agonists, anticholinergic bronchodilators, CNS stimulants
5. Coumarin-type anticoagulants (e.g., warfarin)
6. Symptomatic treatments for acute bronchitis, analgesics (Note: Acetaminophen up to 1.5 g/day taken ≥24 hours before efficacy assessments is permitted)
7. Sedatives
8. Central nervous system depressants
9. Phenytoin
10. Monoamine oxidase (MAO) inhibitors administered within 2 weeks prior to the investigational product or expected to be used during the trial (e.g., antidepressants, antipsychotics, mood stabilizers, anti-Parkinson drugs)

4. Heavy smokers (≥15 cigarettes/day)

* For e-cigarettes, 10 puffs are considered equivalent to one conventional cigarette.

  5. Pregnant or lactating women, or women who are unwilling to use appropriate contraception* or who are planning to become pregnant during the study period.
* Acceptable contraceptive methods include hormonal contraception, intrauterine devices, sterilization of the partner (vasectomy or tubal ligation), or double-barrier methods (e.g., male condom with female diaphragm, sponge, or cervical cap).

  6. Participation in another clinical trial and administration of an investigational drug or device within 4 weeks prior to screening

  7. Any other condition that, in the investigator's judgment, would make the subject unsuitable for participation in this clinical trial

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Bronchitis Severity Score (BSS) total score at Day 4 after dosing | Day 4 after first dose
  The primary efficacy endpoint is the change from baseline in total BSS score at Day 4 after administration of DW5121 compared to DW51211 and DW51212. The BSS is a clinician-rated scale assessing five symptoms of bronchitis (cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea), each scored from 0 (absent) to 4 (very severe), resulting in a total score ranging from 0(no symptoms) to 20(most severe symptoms) where higher scores indicate a worse outcome (more severe bronchitis symptoms).

SECONDARY OUTCOMES:
Change from baseline in Bronchitis Severity Score (BSS) total score at Day 7 after dosing | Day 7 after first dose
  Change from baseline in total BSS score at Day 7 after administration of DW5121 compared to DW51211 and DW51212. The BSS is a clinician-rated scale assessing five symptoms of bronchitis (cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea), each scored from 0 (absent) to 4 (very severe), resulting in a total score ranging from 0(no symptoms) to 20(most severe symptoms), where higher scores indicate a worse outcome (more severe bronchitis symptoms).
Change from baseline in Bronchitis Severity Score (BSS) symptom scores at Days 4 and 7 after dosing | Days 4 and 7 after first dose
  Changes from baseline in individual BSS symptom scores at Days 4 and 7 after administration of DW5121 compared to DW51211 and DW51212. The BSS is a clinician-rated scale assessing five symptoms of bronchitis (cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea), each scored from 0 (absent) to 4 (very severe), resulting in a total score ranging from 0(no symptoms) to 20(most severe symptoms), where higher scores indicate a worse outcome (more severe bronchitis symptoms).
Response rate at Days 4 and 7 after dosing | Days 4 and 7 after first dose
  Response defined as total BSS score ≤3 or a decrease of ≥7 points from baseline at Days 4 and 7 after dosing.
Investigator and patient assessment of overall improvement using a 5-point scale at Days 4 and 7 after dosing | Days 4 and 7 after first dose
  Overall improvement will be assessed separately by the investigator and the patient at Days 4 and 7 after dosing using a protocol-defined 5-point categorical scale. The scale consists of the following categories: 4 (cure), 3 (significant improvement), 2 (improvement), 1 (some improvement), 0 (non-improvement or worsening of symptoms). Higher scores indicate better improvement.
Treatment efficacy rate based on improvement at Days 4 and 7 after dosing | Days 4 and 7 after first dose
  Treatment efficacy defined as "cure" or "significant improvement" based on investigator and patient assessment of overall improvement at Days 4 and 7 after dosing.
Patient satisfaction with treatment using a 5-point scale at Days 4 and 7 after dosing | Days 4 and 7 after first dose
  Patient satisfaction with treatment will be assessed by the patient at Days 4 and 7 after dosing using a protocol-defined 5-point categorical scale. The scale consists of the following categories: 4 (very satisfied), 3 (satisfied), 2 (neutral), 1 (dissatisfied), 0 (very dissatisfied). Higher scores indicate better improvement.
Comparison of Bronchitis Severity Score (BSS) total score changes at Days 4 and 7 after dosing(DW51211 vs DW51212) | Days 4 and 7 after first dose
  Comparison of change from baseline in total BSS score at Days 4 and 7 after administration of DW51211 and DW51212. The BSS is a clinician-rated scale assessing five symptoms of bronchitis (cough, sputum, rales/rhonchi, chest pain during coughing, and dyspnea), each scored from 0 (absent) to 4 (very severe), resulting in a total score ranging from 0(no symptoms) to 20(most severe symptoms), where higher scores indicate a worse outcome (more severe bronchitis symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Jaejeong Shim, Principal Investigator, Principal Investigator — Korea University Guro Hospital
Locations (8):
- South Korea (8):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Yeungnam University Medical Center, Daegu
  - Wonkwang University Hospital, Iksan
  - Kangbuk Samsung Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No